CLINICAL TRIAL: NCT04846738
Title: Comparative Interest of Transcranial Doppler and Quantitative Pupillometry as Neurological Prognostic Factors at 12 Months in Brain Damaged Patients (Stroke or Head Trauma) Admitted to Intensive Care Unit
Brief Title: Transcranial Doppler and Quantitative Pupillometry as Neurological Prognostic Factors in Brain Damaged Patients Admitted to Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN282021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Brain Damage
Keywords: Brain injury; Transcranial Doppler; Quantitative Pupillometry,; neurological prognosis; modified Rankin Score (mRS); Glasgow Outcome Scale Extended (GOS-E)
MeSH Terms: conditions — Brain Injuries | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- brain damaged patients: All major brain damaged patients (stroke or head trauma) admitted to reanimation will be included.
  In the usual practice, they have a Transcranial Doppler and the measurement of the photomotor reflex by quantitative Pupillometry.
  It is planned to collect the simultaneous values of the different parameters during 2,000 measurements.
  The data will be collected retrospectively from 01/12/2020, and prospectively from 01/04/2021.
  Interventions: Device: Transcranial Doppler; Device: Pupillometry.

INTERVENTIONS:
Device: Transcranial Doppler — This device measures Mean Systolic Velocity (VMS), Tele-Diastolic Velocity (TDV) and Pulsatility Index (PI),
Device: Pupillometry. — This device measures the photomotor reflex (basic pupil diameter, percentage of variation, latent and slope of the standard photomotor reflex)
  Other Names: AlgiScan

SUMMARY:
Transcranial Doppler is performed daily in Intensive Care Unit in brain damaged patients. For a few years now, the measurement of the photomotor reflex by quantitative Pupillometry has been routinely performed in Intensive Care Units. The objective of this work is to see if Transcranial Doppler recorded parameters and Pupillary parameters are correlated to the neurological prognosis evaluated at 9 months by the Modified Rankin Score (mRS) and the Glasgow Outcome Scale Extended (GOS-E).

ELIGIBILITY:
Inclusion Criteria:

* All brain damaged patients (stroke or head trauma)
* Admitted to Intensive Care Unit since December 1, 2020

Exclusion Criteria:

* Refusal by the patient or his/her legal representative.
* Benefiting from legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All brain damaged patients (stroke or head trauma), admitted to Intensive Care Unit since December 1, 2020
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score (mRS) (0-5) | Year: 1
  Modified Rankin Score (mRS) measures the degree of disability following a stroke in a patient (level 0 for patients with no symptoms to level 5 for patients with major disability and total dependency)..
Glasgow Outcome Scale Extended (GOS-E) (1-8) | Year: 1
  Glasgow Outcome Scale Extended (GOS-E) measure the impact of brain injured (minimum at 1 (Dead) and maximum at 8 (Upper Good Recovery).

SECONDARY OUTCOMES:
Mean Systolic Velocity (VMS) | At inclusion
  Measured by Transcranial Doppler right and left.
Intra-Cranial Pressure (ICP) | At inclusion
  Collect on medical file.
Pulsatility Index (PI) | At inclusion
  Measured by Transcranial Doppler right and left.
Tele-Diastolic Velocity (TDV) | At inclusion
  Measured by Transcranial Doppler right and left.
Basic pupil diameter | At inclusion
  Measured by Pupillometry right and left
Percentage of variation of the pupil diameter | At inclusion
  Measured by Pupillometry right and left
Latent and slope of the standard photomotor reflex | At inclusion
  Measured by Pupillometry right and left
Tissue Partial Oxygen Pressure (PtiO2) | At inclusion
  Collect on medical file.
Bispectral Index (BIS) | At inclusion
  Collect on medical file. BIS is a reflection of the depth of hypnosis
Richmond Agitation-Sedation Scale (RASS) | At inclusion
  Richmond Agitation-Sedation Scale (RASS) is a symmetrical rating, with positive values for agitation and negative values for the level of consciousness around a point 0 corresponding to a calm and awake patient.
  Collect on medical file.
Heart rate | At inclusion
  Collect on medical file.
Blood pressure | At inclusion
  Collect on medical file.
Natremia (mmol/l) | At inclusion
  Collect on medical file.
Glycemia (mmol/l) | At inclusion
  Collect on medical file.

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No